CLINICAL TRIAL: NCT01754844
Title: A Double-blind Placebo-controlled, Randomised, Single Centre, First Time in Man Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Inhaled Doses of AZD7624 in Healthy Subjects
Brief Title: A First Time in Man Study to Asses the Safety and Tolerability of AZD7624 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D2550C00001
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Phase 1; Healthy Volunteers; Single Ascending Dose (SAD); First Time in Man; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — AZD7624

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1-5, single ascending dose AZD7624 (Experimental): Subjects will participate in 1 of 5 groups. In each group 6 subjects will receive AZD7624 and 2 subjects will receive matching placebo.
  Interventions: Drug: AZD7624
- Placebo (Placebo Comparator): Subjects will participate in 1 of 5 groups. In each group 6 subjects will receive AZD7624 and 2 subjects will receive matching placebo.
  Interventions: Drug: Placebo to match

INTERVENTIONS:
Drug: AZD7624 — Single dose inhaled IMP via a nebulizer
  Arms: Group 1-5, single ascending dose AZD7624
Drug: Placebo to match — Single dose inhaled Placebo via a nebulizer
  Arms: Placebo

SUMMARY:
This is a First in Human study to assess the safety and tolerability of AZD7624, following inhaled administration of single ascending doses in healthy male volunteers and female volunteers of non-child bearing potential. Pharmacokinetics (what the body does to the drug) and pharmacodynamic (what the drug does to the body) parameters will be also assessed as secondary objectives.

DETAILED DESCRIPTION:
A Double-blind Placebo-controlled, Randomised, Single centre, First Time in Man Study to evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Inhaled Doses of AZD7624 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects aged 18 to 55 years
* Able to inhale from the SPIRA nebuliser according to the provided instructions
* Females must have a negative pregnancy test at screening and on admission (Day 1) to the CPU, must not be lactating and must be of non-childbearing potential.
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive and weighing at least 50 kg and no more than 100 kg inclusive.
* FEV1 >80% of the predicted normal value.

Exclusion Criteria:

* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7624
* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or family history of muscle diseases
* Known or suspected history of drug abuse as judged by the Investigator
* Use of any prescribed or non-prescribed medication including antacids, analgesics other than paracetamol/acetaminophen, herbal remedies, vitamins (excluding routine vitamins but including megadose [intake of 20 to 600 times the recommended daily dose])

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, body temperature, ECGs, clinical laboratory safety tests and spirometry) | up to 55 days.

SECONDARY OUTCOMES:
Pharmacokinetics of AZD7624 and assess dose proportionality of the pharmacokinetics following single ascending doses of AZD7624 by assessment of Cmax, t1/2, AUC and CL/F. | Day 1 pre-dose, 5min, 15min, 30min, 1h, 2h, 4h, 6h, 9h,12h, 18h, 24h, 36h, 48h, 56h post dose
Pharmacokinetics of single doses of AZD7624 using the following urine PK parameters: Ae and CLR | Day 1: during 0-6, 6-12, 12-24 and 24-48 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Lindgren, MD, Study Director — AstraZeneca Research and Development SE-431 83 Molndal Sweden; Darren G Wilbraham, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital 6 Newcomen St London SE1 1YR
Locations (1):
- Research Site, London, United Kingdom